CLINICAL TRIAL: NCT05221112
Title: Effects of PNF Patterns Training on Trunk Balance, and Gait in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0218
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Stroke, Ischemic
Keywords: stroke; Gait Disorder; Balance; Disorder,
MeSH Terms: conditions — Ischemic Stroke; Stroke; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: total 30 subjects will be randomly assigned to the experiment group (diagonal pattern training) and the control group (single plane training).Diagonal pattern training will be modified with proprioceptive neuromuscular facilitation technique's chopping and lifting pattern to create 10 movements.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diagonal pattern training (Experimental): diagonal pattern training group will involve performance of proprioceptive neuromuscular facilitation technique's chopping and lifting pattern to create 10 movements.
  Interventions: Other: diagonal pattern training
- control group (Active Comparator): in control group patients will perform movements in single plane
  Interventions: Other: single plane training

INTERVENTIONS:
Other: diagonal pattern training — patients will receive proprioceptive neuromuscular facilitation technique's chopping and lifting pattern to create 10 movements.
  Arms: diagonal pattern training
Other: single plane training — patients will receive single plane training of proprioceptive neuromuscular facilitation in control group
  Arms: control group

SUMMARY:
To determine the effects of PNF patterns Training on trunk balance and gait in chronic stroke patients.

DETAILED DESCRIPTION:
This study will be conducted to investigate the effects of PNF patterns training on the trunk control, balance, and gait ability of chronic stroke patients. Data will be collected from stroke patients from Government Mian Munshi hospital (DHQ) and Riphah Rehabilitation center. A consecutive sampling technique will be use which is based on 6 months' time period. TIS (Trunk Impairment Scale), BBS (Berg Balance Scale), 10 MWT (Meter Walk Test) will be used as a tool to collect the data. SPSS 21 version will be used for data entry and analysis.

This study will provide the effects of PNF patterns training on the trunk control, balance, and gait ability in chronic stroke patients. All possible patients will be taken using random sampling. Single plane training and diagonal pattern training will use. The subjects will randomly assign to the experiment group (diagonal pattern training) and the control group (single plane training). Diagonal pattern training will modified with proprioceptive neuromuscular facilitation technique's chopping and lifting pattern to create 10 movements.

Informed consent will be taken from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients whose onset of stroke was at least 6 months to two years
* Ability to maintain an independent standing posture for 30s, ability to walk 30m alone indoor.
* Patient with the ability to communicate enough and to understand oral instructions given by the therapist.
* Patients who were not using assistive devices
* Patients receiving drug therapy of internal medicine for the alleviation of spasticity.

Exclusion Criteria:

* Unconscious patients.
* Patients undergone Spine surgery.
* Patients with Hemi neglect.
* Sensory ataxia or cerebellar ataxia.
* Coronary heart disease (CHD) or peripheral arterial disease (PAD).
* Cardio respiratory problems.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale | Six months
  This test is used to assess balance and function of trunk in stroke patients
Berg Balance Scale | Six months
  To assess whole body balance
10 Meter Walk Test | Six months
  To assess dynamic mobility

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Criekinge T, Truijen S, Schroder J, Maebe Z, Blanckaert K, van der Waal C, Vink M, Saeys W. The effectiveness of trunk training on trunk control, sitting and standing balance and mobility post-stroke: a systematic review and meta-analysis. Clin Rehabil. 2019 Jun;33(6):992-1002. doi: 10.1177/0269215519830159. Epub 2019 Feb 22. PMID 30791703
- [Background] Zhu Z, Cui L, Yin M, Yu Y, Zhou X, Wang H, Yan H. Hydrotherapy vs. conventional land-based exercise for improving walking and balance after stroke: a randomized controlled trial. Clin Rehabil. 2016 Jun;30(6):587-93. doi: 10.1177/0269215515593392. Epub 2015 Jun 30. PMID 26130657
- [Background] Van Criekinge T, Saeys W, Hallemans A, Velghe S, Viskens PJ, Vereeck L, De Hertogh W, Truijen S. Trunk biomechanics during hemiplegic gait after stroke: A systematic review. Gait Posture. 2017 May;54:133-143. doi: 10.1016/j.gaitpost.2017.03.004. Epub 2017 Mar 4. PMID 28288334
- [Background] Dubey L, Karthikbabu S. Trunk proprioceptive neuromuscular facilitation influences pulmonary function and respiratory muscle strength in a patient with pontine bleed. Neurol India. 2017 Jan-Feb;65(1):183-184. doi: 10.4103/0028-3886.198193. No abstract available. PMID 28084270